CLINICAL TRIAL: NCT07116876
Title: An Open-Label Trial to Assess the Clinical Effectiveness of Matrion Decellularized Placental Membrane Versus Conventional Wound Management in Subjects With Diabetic Foot Ulcers
Brief Title: Matrion Decellularized Placental Membrane Versus Conventional Wound Management in Subjects With Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-24-002
Record Dates: First submitted 2025-08-07; First posted 2025-08-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer (DFU); Lower Extremity
Keywords: diabetic foot ulcer; placental membrane; lower extremity wound; decellularized placental membrane; foot diseases; foot ulcer; conventional wound management
MeSH Terms: conditions — Diabetic Foot; Foot Diseases; Foot Ulcer | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: The study is a post market, multicenter, randomized, open-label trial designed to evaluate the treatment response of Matrion compared to Conventional Wound Management on the wound healing rate of diabetic foot ulcers. Subjects from each clinical site will be evaluated using protocol-specific eligibility criteria to determine who qualifies for study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: (Other): Matrion
  Interventions: Other: Graft Application
- Arm 2 (Other): Conventional Wound Management
  Interventions: Other: Wound Dressing Material

INTERVENTIONS:
Other: Graft Application — Place the graft on the debrided DFU and secure. Follow with conventional care wound management (dressings and off-loading). Product may be applied weekly.
  Other Names: Matrion
  Arms: Arm 1:
Other: Wound Dressing Material — The wound will be debrided and undergo a moist-wound therapy and will be covered with a gauze that is appropriate for the type of wound (moist or dry). Dressings will cover each wound wound for at least 5 days, but no more than 9 days, (7 days +/- 2 days) until the next study visit. Off-loading of the wound is required.
  Arms: Arm 2

SUMMARY:
This study will evaluate Matrion™ (LifeNet Health, Inc., Virginia Beach, VA), a placental membrane product, as a treatment for diabetic foot ulcers compared to conventional wound care. Matrion is derived from donated human birth tissue and includes both the amniotic and chorionic layers, along with the trophoblast layer. It is minimally processed using a proprietary decellularization method and terminally sterilized to ensure the membrane is acellular and sterile, making it suitable for surgical applications.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible to participate in this study, a subject must meet the inclusion criteria listed below:

1. Be male or female and aged between 21 and 80 years at the time of informed consent
2. Have a diagnosis of Type I or Type II diabetes as defined by the American Diabetes Association and have been on a stable anti-diabetic treatment regimen for at least 30 days before the baseline visit.
3. Have full-thickness wound of the lower extremity, below the ankle
4. Have a single target ulcer
5. Have a wound with an area greater than or equal to 1cm2 and less than 25 cm2 with a depth less than or equal to 9 mm
6. Have a diabetic foot ulcer that has been present for at least 30 days with a Wagner Classification Grade 1 or 2:

   * Grade 1: superficial diabetic ulcer involving the full skin thickness but not underlying tissues
   * Grade 2: ulcer extension involving ligament, tendon, joint capsule, or fascia, without presence of abscess or osteomyelitis
7. Have an absence of infection based on Infectious Disease Society of America criteria (assessed at BOTH Screening/Visit 1 and Baseline/Visit 2)
8. Have an adequate circulation to the affected lower extremity, defined as at least one of the criteria within the previous 60 days:

   * Transcutaneous oxygen measurement at the dorsum of the foot greater or equal to 30 mm Hg
   * Ankle-brachial index (ABI) ranging from 0.8 to 1.2
   * At least biphasic Doppler arterial waveforms at the dorsalis pedis and posterior tibial arteries
9. Have the ability to comply with off-loading and dressing change requirements
10. Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an institutional review board (IRB), and agree to abide by the study restrictions and return to the site for the required assessments
11. Have provided written authorization for use and disclosure of protected health information
12. Have a life expectancy of greater than 6 months

Exclusion Criteria:

To be eligible for entry into the study, the subject must not meet any of the exclusion criteria listed below:

1. Be pregnant or lactating
2. Subjects with a target wound <30 days old at Screening whose wound area has decreased in size ≥50% between the Screening and Baseline Visits (assessed at Baseline/Visit 2)
3. Have a circulating hemoglobin A1c exceeding 12% within 90 days of the Screening Visit (assessed at Screening/Visit 1 for subjects with labs collected <30 days of screening; assessed at Baseline/Visit 2 for subjects with labs collected at screening)
4. Have a serum creatinine concentration of 3.0 mg/dL or greater within 30 days prior to screening (assessed at Screening/Visit 1 for subjects with labs collected <30 days of screening; assessed at Baseline/Visit 2 for subjects with labs collected at screening)
5. Have a sensitivity to either of the following antibiotics: lincomycin, gentamicin, polymyxin B, or vancomycin
6. Have a sensitivity to polysorbate 20, N-lauroyl sarcosinate, benzonase or glycerol
7. Have the wound treated with biomedical or topical growth factors within the previous 30 days before the Screening Visit
8. Need for any additional concomitant dressing material other than the ones approved for this study
9. Have clinical signs of an infection at the study ulcer site (assessed at BOTH Screening/Visit 1 and Baseline/Visit 2)
10. Have the inability to tolerate an off-loading boot
11. Have a known or suspected disease of the immune system
12. Have an active or untreated malignancy or active, uncontrolled connective tissue disease
13. Had a treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 30 days before the Baseline Visit
14. Have presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement (assessed at Baseline/Visit 2)
15. Has undergone a revascularization procedure aimed at increasing blood flow in the treatment target limb less than 4 weeks before the Baseline Visit
16. Have serum aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels greater than three times the normal upper limit within 30 days prior to screening (assessed at Screening/Visit 1 if subject had labs collected <30 days of screening; assessed at Baseline/Visit 2 if subject had labs collected at screening)
17. Have active Charcot disease
18. Have undergone treatment with a living skin equivalent within the last 4 weeks before screening
19. Have ongoing evidence of peripheral vascular disease, including greater than one nonpalpable pulse on either foot
20. Have the presence of any condition that in the opinion of the investigator places the subject at undue risk or potentially jeopardizes the quality of the data to be generated

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 12 Weeks
  Proportion of diabetic foot ulcers that have achieved complete wound closure

SECONDARY OUTCOMES:
Speed of Wound Closure | 12 weeks
  Time to wound closure measured from the baseline visit to the termination visit
Change in Wound Area | 12 weeks
  Change in wound area over time
Assessment of Wound Closure Rates in Study Participants | 12 weeks
  Number of subjects with a healed wound
Infection | 12 weeks
  Rate of wound infection
Reoccurrence | 14 weeks
  Rate of re-occurrence of wound during follow-up period
Grafts Used | 12 weeks
  Average number of Matrion grafts used per subject
Incidence of Treatment Emergent Adverse Events | 12 weeks
  Collection of adverse events, including changes in vital signs, ABI, and physical exams

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Compass Medical Research Center, Tucson, Arizona
  - Bay Area Foot Care, Castro Valley, California
  - Limb Preservaion Platform, Inc., Fresno, California
  - Center for Clinical Research, Inc, San Francisco, California
  - Bay Area Foot Care, San Francisco, California
  - ILD Research Center, Vista, California
  - Humanity Clinical Research, Corp, Aventura, Florida
  - South Florida Podiatry, Deerfield Beach, Florida
  - Dinamo Research & Diagnostic Center, LLC, Hialeah, Florida
  - Doctors Research Network, Inc., Miami, Florida
  - Independent Clinical Research, Decatur, Illinois
  - Independent Clinical Research, LLC, Springfield, Illinois
  - US Foot and Ankle Specialists, Raleigh, North Carolina
  - Foot and Ankle Institute of the Carolinas, Rocky Mount, North Carolina
  - Olympus Clinical Research, Katy, Texas
  - Element Research Group, San Antonio, Texas
  - Olympus-Alcanza, Sugar Land, Texas
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No